CLINICAL TRIAL: NCT01173770
Title: A Double-Blind Randomized, Placebo-Controlled, Dose Escalating Study to Assess The Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single and Multiple Doses of ADC3680B Administered Orally to Healthy Volunteers and to Investigate Food Effects on Pharmacokinetics After Single Oral Doses of ADC3680B
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of ADC3680B in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pulmagen Therapeutics (Industry)
Responsible Party: Dr Salvatore Febbraro, Simbec Research Limited
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ADC3680-01
Record Dates: First submitted 2010-07-29; First posted 2010-08-02 (Estimated); Last update posted 2011-02-02 (Estimated); Status verified 2010-07

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Cohort 1: ADC3680B vs. Placebo (Experimental)
  Interventions: Drug: ADC3680B
- Cohort 2: ADC3680B vs. Placebo (Experimental)
  Interventions: Drug: ADC3680B
- Cohort 3: ADC3680B vs Placebo (Experimental)
  Interventions: Drug: ADC3680B
- Cohort 4: ADC3680B vs. Placebo (Experimental)
  Interventions: Drug: ADC3680B
- Cohort 5: ADC3680B vs. Placebo (Experimental)
  Interventions: Drug: ADC3680B
- Cohort 6: ADC3680B (Experimental)
  Interventions: Drug: ADC3680B

INTERVENTIONS:
Drug: ADC3680B — Escalating single doses ADC3680B or Placebo over 5 study periods
  Arms: Cohort 1: ADC3680B vs. Placebo; Cohort 2: ADC3680B vs. Placebo
Drug: ADC3680B — ADC3680B or Placebo for 7 days
  Arms: Cohort 3: ADC3680B vs Placebo; Cohort 4: ADC3680B vs. Placebo; Cohort 5: ADC3680B vs. Placebo
Drug: ADC3680B — Single doses ADC3680B over 2 study periods under fasted and fed conditions
  Arms: Cohort 6: ADC3680B

SUMMARY:
This is a First-In-Man study designed to examine the safety, tolerability, pharmacokinetics and functional activity of ADC3680B after single and multiple doses in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects between the ages of 18 and 55 years
* Body Mass Index (BMI) of 18 to 30 kg/m2
* Signed and dated written informed consent prior to admission into the study
* Willing and able to comply with the requirements of the protocol and available to complete the study

Exclusion Criteria:

* Evidence of history of any clinically significant medical disorder
* History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2010-07; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of single doses of ADC3680B determined by adverse event reporting, clinical laboratory tests, vital signs and ECGs | 2 days
Safety and tolerability of multiple doses of ADC3680B determined by adverse event reporting, clinical laboratory tests, vital signs and ECGs | 8 days

SECONDARY OUTCOMES:
Single dose pharmacokinetics of ADC3680B | 2 days
Multiple dose pharmacokinetic of ADC3680B | 8 days
Pharmacokinetics of ADC3680B under fasted and fed conditions | 2 days
Eosinophil shape change in response to stimulation with PGD2 in whole blood ex vivo | Pre-dose and up to 48 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Febbraro, Principal Investigator — Simbec Research
Locations (1):
- Simbec, Merthyr Tydfil, United Kingdom